CLINICAL TRIAL: NCT03353272
Title: The Influence of a Cognitive Behavioral Approach on Changing Patient Expectations in Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00088013
Record Dates: First submitted 2017-11-21; First posted 2017-11-27 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2022-11

CONDITIONS: Rotator Cuff Impingement Syndrome; Rotator Cuff Injury; Shoulder Pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impairment Based Treatment (No Intervention): an impairment-based conservative intervention that has been created by compiling the evidence associated with established, effective treatment interventions for rotator cuff related shoulder pain.
- Impairment Based Treatment PLUS PEERC (Experimental): Participants assigned to the impairment-based care plus PEERC condition will also receive the PEERC protocol. This protocol, informed by principles of CBT, involves three components: 1) engagement, 2) education and 3) cognitive restructuring and behavioral activation. A health coach who is responsible for engaging patients, educating them about pain modulatory mechanisms, and reinforcing cognitive and behavioral coping skills, will deliver the PEERC protocol.
  Interventions: Behavioral: Patient Engagement Education and Restructuring of Cognitions

INTERVENTIONS:
Behavioral: Patient Engagement Education and Restructuring of Cognitions — This protocol, informed by principles of CBT, involves three components: 1) engagement, 2) education and 3) cognitive restructuring and behavioral activation. A health coach who is responsible for engaging patients, educating them about pain modulatory mechanisms, and reinforcing cognitive and behavioral coping skills, will deliver the PEERC protocol.
  Arms: Impairment Based Treatment PLUS PEERC

SUMMARY:
Background: Despite similar treatment outcomes for surgery or conservative care, the number of surgeries for the care of rotator cuff (RTC) related shoulder pain has increased. With the increase in surgery, there is an increased risk of harms, increased costs, and high re-tear rates. Patient expectations are beliefs or attitudes that include pre-treatment thoughts and beliefs regarding the need for specific treatment methods and the timing and intensity of these methods. Brief interventions designed to alter and enhance treatment expectations for conservative care and have been shown to improve patient expectations, but to date, no studies have explored whether such interventions can influence patient decisions to pursue surgical care. The investigators propose a comprehensive intervention that involves Patient Engagement Education, and Restructuring of Cognitions (PEERC) that is designed to change expectations, will reduce the likelihood that patients will choose to have shoulder surgery and improve functional outcomes. The cognitive behavioral therapy (CBT) approaches that form the core of our PEERC protocol are patient-centered and are designed to empower the patient in their own recovery process.

Purpose/Aims: To examine the effect of the PEERC protocol on the decision to have surgery (primary), and improve global well-being, pain catastrophizing, pain, functional outcomes, and follow up expectations (secondary).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70
* A rotator cuff related shoulder pain diagnosis
* A mobile or land-line telephone
* Ability to read and write English for completion of the self-report forms.

Exclusion Criteria:

* The investigators will exclude patients who have received or are scheduled for a surgical intervention for their shoulder condition
* Demonstrate any evidence of cervicogenic pain and/or radiculopathy from cervical origin
* Who demonstrate symptoms consistent with thoracic outlet syndrome
* The investigators will also exclude individuals who are undergoing treatment for a serious psychological disorder (e.g., severe depression, psychosis).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Pursuance of Surgical Intervention | 6 Months
  The subject will be questioned if, after physical therapy, he or she will pursue surgery to address continued shoulder pain.

SECONDARY OUTCOMES:
Change in Pain | Baseline, 6 weeks, Discharge (estimated 3 months)
  Numeric Pain Scale- The NRS for pain is scaled from 0 to 10 (11 point scale) and is based on pain intensity. Overall pain intensity will be queried where 0/10 represents no pain and 10/10 represents the worst pain possible.
Change in GRoC - Global rate of change | 6 weeks, Discharge (estimated 3 months)
  The Global Rating of Change (GRoC) asks patients to report their global rating of change (GROC) relative to physical function, using a 7-point ordinal scale (where -7 much worse and +7 much better).
Change in SPADI - Shoulder Pain and Disability Index | Baseline, 6 weeks, Discharge (estimated 3 months)
  The SPADI contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability
Change in MODEMS | Baseline, 3 weeks, 6 weeks, Discharge (estimated 3 months)
  The MODEMS patient expectation scale has been used by a number of studies and has shown validity in predicting outcomes in conservative and surgical interventions. As we previously stated, the instrument is a Likert-based scoring tool with a mean score of 5 out of 5 (indicating high expectations of positive outcomes) and a mean score of 1 out of 5 (indicating very poor expectations of positive outcomes)30
Change in TEGNER | Baseline, Discharge (estimated 3 months)
  The Tegner Activity Scale measures the patient's perspective of function and activity as a numerical value between 0 (complete disability) to 10 (elite athletics)
OSPRO 10 - Optimal Screening for Prediction of Referral and Outcome | Baseline
  Optimal Screening for Prediction of Referral and Outcome-10. The OSPRO is a review-of-systems screening tool that includes constructs associated with comorbidities, negative mood, quality of life, pain, and function
Pain Catastrophizing Scale | Baseline
  The Pain Catastrophizing Scale (PCS) assesses the extent of catastrophic thinking according to 3 components: rumination, magnification, and helplessness. It is a 13-item scale
SANE - Single Assessment Numeric Evaluation | 6 months
  The Single Assessment Numeric Evaluation (SANE) is a patient reported outcome measure utilized to rate the patient's perceived level of function
Overall Satisfaction with Care | 6 months
  Patients will be asked to rate their satisfaction of care as "excellent" "good" "fair" or "poor"

CONTACTS AND LOCATIONS:
Overall Officials: Chad E Cook, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Sports Science Institute, Durham, North Carolina, United States

REFERENCES:
- [Derived] Myers H, Keefe FJ, George SZ, Kennedy J, Lake AD, Martinez C, Cook CE. Effect of a Patient Engagement, Education, and Restructuring of Cognitions (PEERC) approach on conservative care in rotator cuff related shoulder pain treatment: a randomized control trial. BMC Musculoskelet Disord. 2023 Dec 1;24(1):930. doi: 10.1186/s12891-023-07044-y. PMID 38041042
- [Derived] Myers H, Keefe F, George SZ, Kennedy J, Lake AD, Martinez C, Cook C. The influence of a cognitive behavioural approach on changing patient expectations for conservative care in shoulder pain treatment: a protocol for a pragmatic randomized controlled trial. BMC Musculoskelet Disord. 2021 Aug 24;22(1):727. doi: 10.1186/s12891-021-04588-9. PMID 34429074